CLINICAL TRIAL: NCT04757948
Title: Acupuncture vs TENS for Gag Reflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew Shubov, MD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#18-000473
Record Dates: First submitted 2021-02-03; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Gagging
Keywords: acupuncture; TENS; acupressure; acupoint; gag
MeSH Terms: conditions — Gagging | interventions — Acupuncture Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Masking of the participant:
  The subject is randomized to one of three groups: 1: acupuncture, 2: TENS, and 3: sham-TENS. While those assigned to the acupuncture group are aware of their group assignment, groups 2 and 3 receive an identical TENS pad placement. A sham-TENS unit is used with disconnected wires to provide a blinking light without an electrical signal. Participants are advised that that the sensation of electrical tingling is not necessary.
  Masking of the examiner:
  The acupuncture or TENS/sham/TENS is performed by one examiner. A second examiner will enter the room to perform the gag reflex measurement, both before and after the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Acupuncture (Experimental): Sterile needles are inserted into acupuncture points P-6 and St-36 bilaterally and retained for a total of 20 minutes. Halfway through the treatment, the needles are manipulated in order to re-create the acupuncture sensation. The needles are removed after 20 minutes of treatment prior to the second gag measurement.
  Interventions: Procedure: Acupuncture
- TENS (Experimental): Gel pads are affixed to the acupuncture points P-6 and St-36, bilaterally. The amplitude of the TENS device will be gradually increased up to a maximum setting of 8/10, with the subject asked to notify the examiner as soon as any sensation is noticed. Once a gentle buzzing sensation is noticed, the amplitude will be reduced slightly for comfort and then the device will remain for the duration of 20 minutes. The pads are then removed prior to the second gag reflex measurement.
  Interventions: Device: TENS
- Sham-TENS (Placebo Comparator): For the sham-TENS group, the protocol is identical to the TENS group, however the electrical wires have been severed and re-attached in the control unit. As such, the unit will flash a light but there will be no current delivered. The subject is told that no sensation is required. The amplitude will be turned up to a maximum setting of 8/10 and left there for 20 minutes, then the device turned off and pads removed.
  Interventions: Device: Sham-TENS

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture of acupoints P-6 and St-36
  Arms: Acupuncture
Device: TENS — TENS of acupoints P-6 and St-36
  Arms: TENS
Device: Sham-TENS — Sham-TENS of acupoints P-6 and St-36
  Arms: Sham-TENS

SUMMARY:
This study examines if acupuncture or TENS of P-6 and St-36 acupoints has a measurable effect on gag tolerance.

DETAILED DESCRIPTION:
The gag reflex is a normal protective mechanism, and portion of the population has an exaggerated reflex that can present major problems in dentistry as well as endoscopy. Early studies with acupuncture have been promising, but these studies are limited as has not been a way to objectively measure the response to gag reflex. Recent work by Drs. Karibe and Goddard has determined a novel way of measuring gag reflex in healthy subjects, which makes it possible to study the effects of an intervention on gag reflex.

Acupuncture has been demonstrated to be effective for treating gag reflex, but this effect has not been objectively demonstrated using this novel method. As such, this study investigates the effect of acupuncture against placebo on gag reflex. Practically speaking, these findings are unlikely to be of high value since the availability of acupuncturists at dental offices is limited. For this reason, the investigators added a third arm to evaluate the use of a transcutaneous electrical nerve stimulator (TENS) device on the same acupuncture points as a treatment intervention to see if this is non-inferior to acupuncture. TENS is an FDA regulated treatment for the treatment of pain, and has been 510K cleared for other uses including nausea. The placebo arm uses a TENS device that has the wire severed, so that the light will continue to blink but no current will be applied.

60 total subjects will be recruited and randomized into one of these three groups: acupuncture, TENS and Sham-TENS.

Passive EKG readings will be collected using the FirstBeat Bodyguard 2, which is a 2-lead EKG device that the subject will wear during the study. This is to later evaluate vagal tone by analyzing the spectral analysis of heart rate variability.

Once this device is affixed to the front of the patient's chest, the gag reflex will be measured. The subject will then undergo the appropriate treatment (acupuncture, TENS or Sham-TENS for a total of 20 minutes, with a subsequent gag reflex measurement. The subject will then rest for at least 5 minutes at the end of the study to collect final EKG data, then given a gift card for her time.

It is the hypothesis of the investigators that the treatments will increase gag tolerance in the following stepwise manner: Sham-TENS < TENS < Acupuncture

ELIGIBILITY:
Inclusion Criteria:

* English Speaking

Exclusion Criteria:

* bleeding dyscrasias
* severe needlephobia
* pacemaker or other implanted electrical device

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Insertion length | immediately after procedure
  A standard saliva ejector with a stopper made of heavy-body addition silicone impression putties is inserted into the participants' mouth at the maxillary central incisor, and gradually guided down the participant's throat along the palate. The participants are asked to inform the examiner when their maximum tolerance has been reached by pushing a button that beeps. The examiner then stopped inserting the saliva ejector, remove it, and measure the insertion distance of the saliva ejector from the maxillary central incisor using digital calipers. This distance is recorded as an index of the gag reflex.
Severity of gag reflex | immediately after procedure
  Subjects are also be asked to report the severity of their gagging on a scale of 1-10, with 1 representing the minimum and 10 representing the maximum

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shubov, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided